CLINICAL TRIAL: NCT03469089
Title: Touchscreen-based Cognitive Tests in Assessment of Ketamine-induced Cognitive Deficits in Healthy Volunteers
Brief Title: Touchscreen-based Cognitive Tests in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: REVISE28347; 2017-004455-22 (EudraCT Number)
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cognitive Symptom; Schizophrenia
Keywords: schizophrenia; cognitive symptom; healthy volunteer; cognitive testing
MeSH Terms: conditions — Neurobehavioral Manifestations; Schizophrenia | interventions — Ketamine; Modafinil

STUDY DESIGN:
Intervention Model Description: All subjects will get each treatment according to balanced latin square design for four treatments with 12 days intervals
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo/placebo (Placebo Comparator): Placebo for ketamine (0.9% NaCl) + Placebo for modafinil (microcrystalline cellulose capsule)
  Interventions: Drug: Placebo for ketamine; Drug: Placebo for modafinil
- Ketamine 0.58/placebo (Experimental): Ketamine (0.23 mg/kg + 0.58 mg/kg/h) + Placebo for modafinil
  Interventions: Drug: Ketamine 0.58; Drug: Placebo for modafinil
- Ketamine 0.58/modafinil (Experimental): Ketamine (0.23 mg/kg + 0.58 mg/kg/h) + Modafinil (200 mg)
  Interventions: Drug: Ketamine 0.58; Drug: Modafinil
- Ketamine 0.31/placebo (Experimental): Ketamine (0.12 mg/kg + 0.31 mg/kg/h) + Placebo for modafinil
  Interventions: Drug: Ketamine 0.31; Drug: Placebo for modafinil

INTERVENTIONS:
Drug: Ketamine 0.58 — Ketamine (0.23 mg/kg bolus + 0.58 mg/kg/h)
  Other Names: Ketalar
  Arms: Ketamine 0.58/modafinil; Ketamine 0.58/placebo
Drug: Ketamine 0.31 — Ketamine (0.12 mg/kg bolus + 0.31 mg/kg/h)
  Other Names: Ketalar
  Arms: Ketamine 0.31/placebo
Drug: Modafinil — Modafinil tablet 100 mg placed in a capsule
  Other Names: Modafinil Orion
  Arms: Ketamine 0.58/modafinil
Drug: Placebo for ketamine — 0.9 % NaCl infusion solution
  Other Names: Placebo
  Arms: Placebo/placebo
Drug: Placebo for modafinil — Placebo capsule for modafinil capsule
  Other Names: Placebo
  Arms: Ketamine 0.31/placebo; Ketamine 0.58/placebo; Placebo/placebo

SUMMARY:
This phase Ib study aims to evaluate applicability of touchscreen-based cognitive test battery for assessment of ketamine-induced schizophrenia-like cognitive deficits in healthy volunteers. Additionally, the study aims to assess whether ketamine-induced cognitive deficits are reversed by modafinil using touchscreen-based test battery for testing of cognition.

DETAILED DESCRIPTION:
Ketamine-induced schizophrenia-like cognitive deficits in healthy volunteers are measured by using touchscreen-based cognitive tests. In addition, the study aims to assess whether ketamine-induced cognitive deficits detected by touchscreen-based cognitive tests are reversed by modafinil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian men aged 20-40 years
* Body weight 50-100 kg
* Body mass index 19-26 kg/cm2
* Normal physical examination including heart rate (HR; 50-90/min) blood pressure (BP; diastolic 65-90 and systolic 110-140) normal haematological and clinical chemistry variables normal ECG as judged by the investigator

Exclusion Criteria:

* Visual disability or red-green color blindness
* History of mental health disorders as determined by self-reported a) physician-determined diagnoses of mental health disorders, except for nicotine and caffeine dependence, or history of suicide attempt; b) medications for mental health disorders
* History of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, or neurological disorder
* History of orthostatic syncope
* History of head injury with sequelae
* First-degree relative with a history of psychosis or epilepsy/seizure disorder or of a condition with risk of seizures
* Current regular medication
* Vaccination 2 weeks prior to study or during the study
* Known or suspected allergy/hypersensitivity to any drug
* History of regular alcohol consumption
* Current substance dependence (excluding nicotine and caffeine).
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day
* Use of any medication or alcohol 24 hours before each study visit
* Education less than high school
* Clinically relevant symptoms of depression, anxiety or sleep disturbances
* Donation of blood within 1 month prior to study
* Participation in any study with an investigational product within 2 months prior to study
* Clinical signs of suicidal or violent behaviour or psychotic symptoms

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Ketamine-induced cognitive deficits | 15-60 min after initiation of ketamine or placebo infusion
  Ketamine-induced cognitive deficits are measured by using the touchscreen cognitive test battery

SECONDARY OUTCOMES:
Effect of modafinil on ketamine-induced cognitive deficits | 15-60 min after initiation of ketamine or placebo infusion
  The effect of modafinil on ketamine-induced cognitive deficits are measured by using the touchscreen cognitive test battery

OTHER OUTCOMES:
Ketamine plasma levels | 14 and 60 min after initiation of ketamine or placebo infusion
  Assessment of ketamine plasma levels
Brain-derived neurotrophic factor serum levels | 14 and 60 min after initiation of ketamine of placebo infusion
  Assessment of Brain-derived neurotrophic factor serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Markus M Forsberg, PhD, Study Director — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Clinical Research Centre, Brain Research Unit, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided